CLINICAL TRIAL: NCT07179536
Title: Optimizing Time to Ambulation After ProGlide Closure of Femoral Access: A Randomized Controlled Trial
Brief Title: Time to Ambulation After ProGlide Closure
Acronym: OPTIMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Hui DONG, professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0906
Record Dates: First submitted 2025-09-16; First posted 2025-09-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Femoral Access Site Closure; Ambulation; Vascular Access Complication; Vascular Access Site Management
Keywords: Femoral access site closure; Vascular closure device; Time to ambulation; Vascular access complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Ambulation (2 hours) (Experimental): Patients instructed to ambulate 2 hours after ProGlide femoral artery closure.
  Interventions: Procedure: Ambulation after ProGlide Closure
- Intermediate Ambulation (6 hours) (Experimental): Patients instructed to ambulate 6 hours after ProGlide femoral artery closure.
  Interventions: Procedure: Ambulation after ProGlide Closure
- Late Ambulation (12 hours) (Experimental): Patients instructed to ambulate 12 hours after femoral access site closure with ProGlide.
  Interventions: Procedure: Ambulation after ProGlide Closure

INTERVENTIONS:
Procedure: Ambulation after ProGlide Closure — Ambulation time after femoral artery access site closure using the ProGlide vascular closure device was assigned to 2 hours, 6 hours, or 12 hours post-procedure.

SUMMARY:
Transradial access has become the standard for coronary procedures due to fewer vascular complications and shorter bed rest, yet transfemoral access remains essential for complex peripheral interventions requiring larger sheaths and stronger support. Vascular closure devices (VCDs), particularly suture-mediated devices such as ProGlide, have improved femoral access by reducing hemostasis time, ambulation delay, and patient discomfort. Although early ambulation after ProGlide closure has been reported, current practice varies widely, and the relationship between ambulation timing and vascular complications remains unclear. This trial aims to evaluate the effect of different ambulation times after ProGlide closure in transfemoral peripheral angiography or intervention, with the goal of identifying the optimal time to ambulation that balances safety and efficiency.

DETAILED DESCRIPTION:
Transradial access has replaced transfemoral access as the mainstream approach for coronary angiography and intervention due to its lower incidence of vascular complications and shorter postoperative bed rest. In non-coronary endovascular interventions, radial access is also an attractive alternative. However, the traditional femoral approach retains irreplaceable advantages: it is easier for puncture and sheath insertion, accommodates sheaths ≥ 8F, allows the delivery of larger stents, provides better guiding catheter support, and reduces procedural difficulty and time.

In recent years, the widespread use of vascular closure devices (VCDs) has further improved the physician and patient experience of femoral access. Compared with manual compression, VCDs significantly reduce hemostasis time, shorten postoperative bed rest, and improve patient comfort and satisfaction. VCDs can be classified into four categories based on the closure mechanism: collagen plug, suture-mediated, disc-based, and metal clip. Although comparative studies among different VCDs are limited, the efficacy and safety of suture-mediated VCDs have been well demonstrated. ProGlide, as a representative of suture-mediated VCDs, is favored for large sheath compatibility, reliable hemostasis, and low vascular complication rates.

Evidence from Aravind Sekhar et al. showed that patients undergoing diagnostic coronary angiography via femoral access could ambulate early after ProGlide closure, which is a key driver for reducing hospitalization time, lowering costs, and improving patient satisfaction. While previous studies have reported the benefit of VCDs in shortening time to ambulation, the determination of ambulation time was largely empirical, ranging from 2 to 12 hours depending on operator experience. Currently, there is a lack of evidence regarding the association between ambulation time and vascular complications at the access site. This study aims to investigate the impact of different ambulation times after ProGlide closure in patients undergoing transfemoral peripheral angiography or endovascular intervention on vascular access site complications, in order to determine the optimal timing for ambulation.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for peripheral angiography or endovascular intervention via transfemoral access.
* Femoral artery puncture site located at the common femoral artery.
* Use of 6-8F vascular sheath.
* Hemostasis achieved with 6F ProGlide closure device (defined as no active bleeding, no hematoma formation, and no ischemia of the punctured limb after closure).
* Preoperative ankle-brachial index (ABI) > 0.9 on both sides.
* Conscious, cooperative, and with normal lower limb mobility.

Exclusion Criteria:

* Undergoing carotid artery intervention.
* Femoral artery diameter < 5 mm, or effective lumen < 5 mm due to plaque burden.
* History of vascular complications at the puncture site.
* Abnormal cardiopulmonary function.
* Intraoperative platelet count < 80 × 10⁹/L, or use of thrombolytic agents.
* Cognitive impairment, uncooperative, or limited lower limb mobility.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Femoral Access Site Vascular Complications | Within 24 hours post-procedure or before hospital discharge (whichever comes first)
  Composite outcome of femoral access site vascular complications, defined as the occurrence of any of the following: (1)Bleeding events classified as BARC type 2 or higher;(2)Hematoma > 5 cm in diameter;(3)Pseudoaneurysm ;(4)Arteriovenous fistula;(5)Femoral artery stenosis or occlusion

SECONDARY OUTCOMES:
Ankle-Brachial Index (ABI) Changes | Before discharge
  Measurement of ABI to assess potential femoral artery stenosis or occlusion at the puncture site
Pain at Access Site (Visual Analog Scale, VAS) | 24 hours post-procedure
  Patient-reported pain score (0-10 scale) at the femoral access site.
Vascular Complications within 30 Days | 30 days post-procedure
  Incidence of late access-site complications, including delayed bleeding, pseudoaneurysm, arteriovenous fistula, or femoral artery stenosis/occlusion requiring clinical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Dong, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China